CLINICAL TRIAL: NCT00902564
Title: Efficacy and Safety of Escitalopram in Patients With Generalized Anxiety Disorder; Open-label, One Arm Postmarketing Study in Russia
Brief Title: Escitalopram in Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: H. Lundbeck A/S, H. Lundbeck A/S
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12132A
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Results first posted 2011-06-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-05

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; GAD; Antidepressant; Anxiolytic
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Escitalopram (Experimental)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Flexible-dosed (5 to 20 mg Oral Tablets Daily)
  Other Names: Cipralex, Lexapro

SUMMARY:
The purpose of this study is to evaluate the effect of escitalopram after 8 weeks of treatment in patients with Generalized Anxiety Disorder (GAD), to evaluate proportion of patients who respond to escitalopram during the treatment period, and to evaluate safety of escitalopram.

DETAILED DESCRIPTION:
The study will be performed in Russia, as an open-label, uncontrolled, one arm trial. The patients will receive escitalopram for 8 weeks. Start and maintenance dosages as well as dose titration will be left to the investigators' decision (5 to 20 mg/day), in accordance with the national Summary of Products Characteristics (SPC).

ELIGIBILITY:
Inclusion Criteria:

* The patient suffers from GAD, diagnosed according to ICD-10 (International Classification of Diseases)
* The patient meets criteria as set out in the national SPC for escitalopram
* The patient is, in the opinion of the investigator, otherwise healthy on the basis of a physical examination, medical history and vital signs

Exclusion Criteria:

* The patient has/has had an alcohol or drug abuse-related disorder, as defined in ICD-10
* The patient has contraindications to escitalopram
* The patient has a history of severe drug allergy or hypersensitivity, or known hypersensitivity to escitalopram
* The patient has a serious illness and/or serious sequelae thereof, including liver or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic, or metabolic disturbance
* The patient is pregnant or breast-feeding
* The patient, if a woman of childbearing potential, is not using adequate contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- RU001, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Started | 30
Completed | 28
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.3 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Hamilton Anxiety Scale (HAMA) [Mean (Standard Deviation); unit: scores on a scale] — The HAMA is a 14-item rating scale designed to assess global anxiety symptoms. Each symptom is rated from 0 (absent) to 4 (severe). The total score of the 14 items ranges from 0 to 56.
  scores on a scale | 31.1 (5.3)
Clinical Global Impression Severity (CGI-S) [Mean (Standard Deviation); unit: scores on a scale] — The CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients).
  scores on a scale | 4.5 (0.6)
Sheehan Disability Scale (SDS) Work [Mean (Standard Deviation); unit: scores on a scale] — The SDS comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scale, on which 0 = normal functioning and 10 = severe functional impairment.
  scores on a scale | 6.8 (1.6)
Sheehan Disability Scale (SDS) Family [Mean (Standard Deviation); unit: scores on a scale] — The SDS comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scale, on which 0 = normal functioning and 10 = severe functional impairment.
  scores on a scale | 6.1 (2.0)
Sheehan Disability Scale (SDS) Social [Mean (Standard Deviation); unit: scores on a scale] — The SDS comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scale, on which 0 = normal functioning and 10 = severe functional impairment.
  scores on a scale | 6.8 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Escitalopram After 8 Weeks of Treatment in Patients With GAD Using the Hamilton Anxiety Scale (HAMA)
Description: The HAMA is a 14-item rating scale designed to assess global anxiety symptoms. Each symptom is rated from 0 (absent) to 4 (severe). The total score of the 14 items ranges from 0 to 56.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Number analyzed (Participants) | 28
scores on a scale | 13.1 (6.2)

2. Secondary Outcome: Effect of Escitalopram After 8 Weeks Using the Clinical Global Impression (CGI-I)
Description: The CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Number analyzed (Participants) | 28
scores on a scale | 1.2 (0.4)

3. Secondary Outcome: Effect of Escitalopram After 8 Weeks Using the Clinical Global Impression (CGI-S)
Description: The CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients).
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Number analyzed (Participants) | 28
scores on a scale | 1.9 (0.7)

4. Secondary Outcome: Percentage of Patients Who Responded to Escitalopram After 8 Weeks of Treatment Using CGI-I <= 2
Description: as for outcome 2
Time Frame: baseline and 8 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Number analyzed (Participants) | 28
percentage of patients | 100

5. Secondary Outcome: Percentage of Patients Who Achieved Remission After 8 Weeks of Treatment Using CGI-S <= 2
Description: as for outcome 3
Time Frame: baseline and 8 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Number analyzed (Participants) | 28
percentage of patients | 85.7

6. Secondary Outcome: Effect of Escitalopram After 8 Weeks Using Sheehan Disability Scale (SDS) Work
Description: The SDS comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scale, on which 0 = normal functioning and 10 = severe functional impairment.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Number analyzed (Participants) | 21
scores on a scale | 2.0 (2.0)

7. Secondary Outcome: Effect of Escitalopram After 8 Weeks Using Sheehan Disability Scale (SDS) Family
Description: as for outcome 6
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Number analyzed (Participants) | 28
scores on a scale | 1.2 (1.9)

8. Secondary Outcome: Effect of Escitalopram After 8 Weeks Using Sheehan Disability Scale (SDS) Social
Description: as for outcome 6
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Number analyzed (Participants) | 28
scores on a scale | 1.7 (2.4)

9. Secondary Outcome: Percentage of Patients Who Responded According to >= 50% Improvement From Baseline to Week 8 in HAMA Total Score
Description: as for outcome 1
Time Frame: baseline and 8 weeks
Population: Observed Cases (OC)
Measure: Number; unit: percentage of patients
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Number analyzed (Participants) | 28
percentage of patients | 67.9

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Escitalopram (5 to 20 mg Oral Tablets Daily)
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 13/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (5 to 20 mg Oral Tablets Daily) (N=30)
Dry mouth (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No results can be made public before appropriate steps by Lundbeck to secure patents and/or intellectual property rights. The Investigator shall send any manuscript and/or public presentation to Lundbeck at least 1 month before submission for publication. If Lundbeck finds matters requiring patents or the like, the Investigator shall delay publication and/or public presentation for an additional 3 months.